CLINICAL TRIAL: NCT06556784
Title: At-home Immersive Virtual Reality Exergames to Reduce Cardiometabolic Risk Among Office Workers: Protocol for a Randomized Controlled Trial
Brief Title: Immersive Virtual Reality Exergames and Office Workers' Cardiometabolic Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University (Other)
Responsible Party: Principal Investigator, Zhao Jing, Associate Researcher, Guangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VRGOWH2024Z
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Exergaming; Metabolic Syndrome
Keywords: Immersive virtual reality; Physical activity; Office workers
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: A 2-armed, single blinded randomized controlled trial (RCT) will be applied to examine the therapeutic effects of at-home immersive virtual reality exergame in this exploratory study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The trial will be conducted in a single-blinded structure, ensuring that all the participants are blinded to treatment or control related information. The experiment coordinators are unblinded and responsible for labelling the groups, allocating experimental equipment and materials, gathering data from participants and clinics, and analyzing all the relationships between and within the two groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-week at-home immersive virtual reality exergame (Experimental): 12-week training of at least 150 minutes per week at-home immersive virtual reality exergame playing with a set device of Meta Quest 2 and maintaining regular eating and working habits without making significant changes.
  Interventions: Behavioral: 12-week at-home immersive virtual reality exergame
- 12-week control in awaiting (No Intervention): Maintaining regular eating and working habits without making significant changes throughout the 12 weeks.

INTERVENTIONS:
Behavioral: 12-week at-home immersive virtual reality exergame — 12-week training of at least 150 minutes per week at-home immersive virtual reality exergame playing with a set device of Meta Quest 2 and maintaining regular eating and working habits without making significant changes.
  Arms: 12-week at-home immersive virtual reality exergame

SUMMARY:
The worldwide increasing of prevalence of non-communicable diseases has grown the recognition of necessity for identifying the modifiable risk in preventing and managing these diseases. While, the office worker, as a representative group of physical inactivity, is exposed to risk factor of metabolic syndrome which is considered as the pathway of non-communicable diseases. This study mainly focuses on the purpose of examining the interventional efficacy of at-home immersive virtual reality exergame on several metabolic syndrome biomarkers among office workers. In addition, it purposes to determine the impacts of at-home immersive virtual reality exergame on lifestyle pattern of office workers. A 2-armed, single blinded randomized controlled trial (RCT) will be applied to examine the therapeutic effects of at-home immersive virtual reality exergame in this exploratory study. 120 Japanese office workers with less than 150 minutes per week of moderate to vigorous sports activities will be recruited by a convenience sample method. They are randomly allocated to two parallel groups, which including an intervention group: 12-week training of at least 150 minutes per week at-home immersive virtual reality exergame playing with a set device of Meta Quest 2, a control group: 12-week of maintaining regular exercise, eating, and working habits without making significant changes. During this 12-week trial, 3 main follow up steps are included at the timelines of 0 week, 6 weeks, 12 weeks. For each follow up, we will collect three types of variables, including major clinical risk factors of metabolic syndrome, lifestyle pattern factors of metabolic syndrome, and demographics (0 week only). To analysis the variance between intervention group and control group, mixed linear model will be applied to understand the efficacy result of this intervention. The variances of metabolic syndrome clinical risk factors between groups would be used to express the therapeutic effects of at-home immersive virtual reality exergame. The changes of lifestyle pattern factors would be applied to show the impacts of at-home immersive virtual reality exergame on lifestyle pattern.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old
* Capable of standing and exercising.
* Having no history of diagnosis of heart disease, cancer, or dementia.
* Being interested in playing with the exergames.
* Willingness of adhering to a 12-week interventional exergame treatment.

Exclusion Criteria:

* Individuals who are already engaged in more than 150 minutes per week of moderate to vigorous activities.
* Individuals with some pharmacological treatments, some surgery (bariatric surgery), and some traditional Chinese medicine.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
High-density lipoprotein cholesterol (HDL-C) | Baseline (0 week), Mid-follow up (6-week), Final follow up (12-week).
  HDL-C concentration less than 35 mg/dl for men (39 mg/dl for women).
Low-density lipoprotein cholesterol (LDL-C) | Baseline (0 week), Mid-follow up (6-week), Final follow up (12-week).
  LDL-C < 160 mg/dl
Impaired fasting glucose | Baseline (0 week), Mid-follow up (6-week), Final follow up (12-week).
  a fasting plasma glucose (FPG) concentration between 6.1 and 6.9 mmol/l.
Triglycerides | Baseline (0 week), Mid-follow up (6-week), Final follow up (12-week).
  Triglycerides concentration > 150 mg/dl.
Hypertension | Baseline (0 week), Mid-follow up (6-week), Final follow up (12-week).
  a Systolic blood pressure > 140 mmHg AND diastolic blood pressure < 90 mmHg.
Body mass index | Baseline (0 week), Mid-follow up (6-week), Final follow up (12-week).
  Weight and height will be combined to report body mass index in kg/m^2.

SECONDARY OUTCOMES:
Exercise time (including exergaming time) | Baseline (0 week, self estimation), Mid-follow up (1-6 week), Final follow up (7-12 week).
  Total minutes of exercise time and exergaming time per week.
Sedentary time | Baseline (0 week, self estimation), Mid-follow up (1-6 week), Final follow up (7-12 week).
  Total minutes of sedentary time per week.

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the IPD.

REFERENCES:
- [Derived] Zhao J, Yasunaga A, Kaczynski AT, Park H, Luo Y, Li J, Shibata A, Ishii K, Yano S, Oka K, Koohsari MJ. At-Home Immersive Virtual Reality Exergames to Reduce Cardiometabolic Risk Among Office Workers: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jan 20;14:e64560. doi: 10.2196/64560. PMID 39832174